CLINICAL TRIAL: NCT02812940
Title: A Single-centre Study of Certican (Everolimus) as Prophylaxis for Graft-versus-Host Disease Following Post-Transplantation Cyclophosphamide After Allogeneic Stem Cell Transplantation
Brief Title: Single-centre Study of Everolimus as GvHD Prophylaxis After Post-Transplantation Cyclophosphamide After Allogeneic SCT
Acronym: OCTET-Ever
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Christoph Scheid, Prof. Dr. Christoph Scheid, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Uni-Koeln 1717
Record Dates: First submitted 2016-06-19; First posted 2016-06-24 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Graft-versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus as part of GvHD prophylaxis after allogeneic SCT (Experimental): Everolimus from day +5 to day +100
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — GvHD prophylaxis
  Other Names: Certican

SUMMARY:
A phase II clinical study to assess the efficacy of short-term everolimus as prophylaxis for Graft-versus-Host disease (GvHD) in addition to post-transplantation cyclophosphamide after allogeneic hematopoietic stem cell transplantation in patients with haematological malignancies

DETAILED DESCRIPTION:
Title of the clinical study: A single-centre study of Certican (everolimus) as Prophylaxis for Graft-versus-Host Disease following Post-Transplantation Cyclophosphamide after Allogeneic Stem Cell Transplantation (OCTET-EVER)

Indication: Patients with haematological malignancies after allogeneic haematopoietic stem cell transplantation with a matched related or unrelated donor following reduced intensity conditioning and post-transplantation cyclophosphamide

Phase: Phase II clinical study

Type of study, study design, methodology: Single centre single arm clinical trial, A'Hern's single stage phase II procedure

Number of subjects: 20 (17 total evaluable)

Primary study objective To assess the efficacy of short-term everolimus as GvHD prophylaxis in addition to post-transplantation cyclophosphamide after allogeneic hematopoietic stem cell transplantation in patients with haematological malignancies and to describe the influence of the modified immunosuppression concept on the incidence and severity of acute GvHD, relapse rates, minimal residual disease, immune reconstitution and chimerism.

Medical condition or disease to be investigated:

• Patients with haematological malignancies after allogeneic haematopoietic stem cell transplantation with a matched related or unrelated donor following reduced intensity conditioning and post-transplantation cyclophosphamide

Name of investigational medicinal product (IMP): Everolimus (Certican®) Investigational medicinal product - dosage and method of administration: 1,5mg per os twice a day (target blood level 5 to 10ng/ml) from day +5 to day +100 after allogeneic stem cell transplantation

Duration of treatment: The treatment will be given from day +5 to day +100 after allogeneic stem cell transplantation. The observation time will last from day +5 to day +130. Incidence of chronic GvHD, overall survival and relapse incidence will be recorded on d+365 and d+720 after transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological malignancies after allogeneic haematopoietic stem cell transplantation with a matched related or unrelated donor following reduced intensity conditioning and post-transplantation cyclophosphamide

Principal inclusion criteria:

• Written informed consent

Exclusion Criteria:

* Known intolerance to everolimus
* Presence or history of Microangiopathy
* Presence of uncontrolled infections
* Severe organ dysfunction defined as:
* Cardiac left ventricular ejection fraction (LVEF) of less than 35%
* Diffusing lung capacity (DLCO) of less than 40%
* Total lung capacity (TLC) of less than 40%
* Forced expiratory volume (FEV1) of less than 40%
* Total bilirubin >3mg/dl
* Creatinine-clearance of less than 40 ml/min
* Pregnancy or breast feeding
* Participation in other experimental drug trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-04; Primary Completion 2019-07 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Incidence of acute GvHD III-IV° until day +100 after allogenic stem cell transplantation | day 100 after transplantation
  GvHD

SECONDARY OUTCOMES:
Incidence of acute GvHD II-IV° until day +100 after allogenic stem cell transplantation | day 100 after transplantation
  GvHD
Incidence of severe chronic GvHD | 720 days after transplantation
  cGvHD
Incidence of overall chronic GvHD | 720 days after transplantation
  cGvHD
Relapse incidence | 720 days after transplantation
  Relapse
Non-relapse mortality | 720 days after transplantation
  NRM
Overall survival | 720 days after transplantation
  OS
Immune reconstitution | day 100 after transplantation
  Number of CD3, CD4, CD8, CD20 and CD56 positive cells in peripheral blood
Engraftment | day 100 after transplantation
  absolute neutrophil count > 500/ul and platelet count > 50.000/ul
Chimerism | day 100 after transplantation
  % donor cells in peripheral blood or bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Christof Scheid, Prof. Dr., Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No